CLINICAL TRIAL: NCT00663247
Title: Mechanistic Randomized Controlled Trial of Mesalazine in Symptomatic Diverticular Disease
Brief Title: Mechanistic Randomized Controlled Trial (RCT) of Mesalazine in Symptomatic Diverticular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07057
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Diverticulosis, Colonic
Keywords: Diverticular disease; Inflammation; Mesalazine
MeSH Terms: conditions — Diverticulosis, Colonic; Diverticular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator): placebo used as control for comparison with active drug
  Interventions: Drug: Placebo
- A (Active Comparator)
  Interventions: Device: Mesalazine

INTERVENTIONS:
Device: Mesalazine — 3 grams daily for 3 months
  Other Names: Salofalk®; 5 ASA
  Arms: A
Drug: Placebo — 3 grams daily for 3 months
  Other Names: Sham medication
  Arms: B

SUMMARY:
Diverticulosis (bulges in the bowel wall) affects two third of the elderly population in the UK. Diverticular disease and its complications are responsible for 68000 hospital admissions and 2000 deaths per year. It commonly produces recurrent short lived abdominal pain, changes in bowel habit and incontinence. The causes of symptoms are not known and the treatments unsatisfactory. Recent studies have found an association between inflammation, alteration of bowel nerves and symptoms. Mesalazine is an anti-inflammatory drug used in inflammatory bowel conditions, such as ulcerative colitis and crohn's disease. We plan to perform a randomized double blind (neither the patients or the doctors known which treatment the patient is taking) placebo (sham medication) controlled trial of mesalazine in symptomatic diverticular disease patients. We anticipate a reduction in the amount of inflammation, bowel nerve changes and symptoms in patients taking mesalazine compare to those taking the placebo.

DETAILED DESCRIPTION:
Diverticular disease affects two thirds of the elderly population in the United Kingdom. Only a small fraction of individuals with diverticulosis develop symptoms, perhaps 1 in 10, for reasons which are not well understood. The symptoms however are quite disabling as we found in a recent survey which indicated that around 36% suffered recurrent abdominal pain. Surprisingly, given the severity of the disability there has been very little research into the factors predicting the development of painful diverticular disease. Recent studies have indicated however that there may be an inflammatory component since the best predictor of recurrent abdominal pain is a previous episode of acute diverticulitis.

Just what initiates an attack of acute diverticulitis is poorly understood but may include the inspissation of fecal material in the diverticulum which then leads to pressure on the lining epithelium and a break down of barrier function. This allows colonic bacteria to enter the lamina propria where they cause acute inflammation, attracting pus cells from the circulating blood and creating micro-abscesses. The resolution of this involves fibrosis and scaring together with muscular hypertrophy which may well lead to secondary motor abnormalities. Patients with symptomatic diverticular disease are known to have higher intraluminal pressures, both at baseline and in response to stimuli such as a meal or prostigmine.

A recent report in which patients admitted with acute diverticulitis were followed for two years found that a very high proportion of such individuals subsequently develop recurrent chronic abdominal pain. Recent work has indicated that this leaves a permanent change in mucosal innervation. Markers of nerve injury including galanin and substance P are upregulated in patients with symptoms as opposed to those without. This is the first time that an objective marker has been shown to distinguish patients on the basis of symptoms.

While acute diverticulitis may be the initiating insult, a chronic low level inflammation may also be required to maintain visceral hypersensitivity. Where detailed quantitative histology has been performed in diverticular disease, some individuals have been identified with a lymphocytic infiltration. In other circumstances, chronic inflammation sensitises mucosal nerves and is associated with visceral hypersensitivity, something which has also been noted in symptomatic diverticular disease.

Whether anti-inflammatory agents could reverse this process is as yet unknown but there are currently available safe and effective treatments for inflammatory bowel disease such as 5 amino-salicylic acid or budesonide which might well be effective and allow further evaluation of the role of low grade inflammation in symptomatic diverticular disease.

This study aims to investigate the inflammatory, neurological and symptomatic effects of mesalazine in diverticular disease.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic diverticular disease with short lived recurrent abdominal pain on 3 or more days a month.
* 18 - 85 years of age.
* Signed informed consent
* Presence of at least one diverticulum in the left colon

Exclusion Criteria:

* Pregnant or lactating women.
* Severe co-morbidity, alcoholism or drug dependence or inability to give informed consent.
* Contraindications to use of Mesalazine as detailed in SmPC.
* Inability to stop NSAIDs (non-steroidal anti-inflammatory agents) or long term antibiotics.
* The use of specific concomitant medications as detailed in the section below.
* Presence of other gastrointestinal inflammatory conditions such as ulcerative colitis, Crohn's disease and Coeliac disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Difference in galanin expression in mucosal nerves from 0 to 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: RC Spiller, Prof, Principal Investigator — Nottingham University Hospital
Locations (1):
- NIHR Biomedical Research Unit, Nottingham University Hospital, Nottingham, Nottinghamshire, United Kingdom